CLINICAL TRIAL: NCT06050330
Title: CD4+ T Cells and S100A7 Epression in Normal and Psoriatic Skin: A Histological and Histochemical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ashrakat Abdelhamid Amin, principle investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-23-09-01MS
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases group (Active Comparator): patients with psoriasis
  Interventions: Diagnostic Test: skin biopsy
- control group (Active Comparator): Healthy
  Interventions: Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: skin biopsy — Paraffin sections,5 Um thick will be prepared from the skin samples and will be analyzed for light microscopy

SUMMARY:
Psoriasis is one of the commonest and most researched chronic immune-mediated inflammatory skin disorders that affects approximately 1-3% of the population worldwide and significantly impairs patients' quality of life. The most common form is plaque psoriasis, which makes up about 90% of cases, which primarily manifests as sharply demarcated, erythematous, scaly plaques, which can involve any part of the skin but most commonly the extensor surfaces (such as the elbows and knees) and the scalp. Apart from plaque psoriasis, there are also other clinical forms, such as guttate psoriasis (particularly common in children after strep throat infections), and pustular psoriasis (one of the most severe varieties of psoriasis, in which the spreading of pustules is generalized, with epidermal fulfillment and a severe general condition).

This disease is characterized by alternating severity and remission of disease symptoms, which include the formation of skin lesions of varying severity. The psoriasis area and severity index (PASI) is a widely used instrument in psoriasis trials that assesses and grades the severity of psoriatic lesions and the patient's response to treatment. It produces a numeric score ranging from 0 to 72. In general, a score of 5 to 10 is considered moderate disease, and a score over 10 is considered severe.

A series of basic and clinical studies have shown that psoriasis is mediated by components of both the innate and adaptive immune systems. The crosstalk between keratinocytes and various immune cells, especially helper T cells, plays a central role in the progression of psoriasis. Psoriasis is caused by chronic interaction between keratinocytes and activated immune cells. Numerous studies have established that hyperproliferation and abnormal differentiation of keratinocytes is a secondary phenomenon induced by immune activation. This "immune" hypothesis, is mainly based on dendritic cell (DC) and T cell pathogenic functions.The abnormal expression of S100A7 as a part of innate immunity in psoriasis vulgaris has been confirmed. S100 proteins are being discussed not only as potential biomarkers as well as new therapeutic targets through inhibition of S100 protein expression, targeted degradation, and antibody-mediated binding of S100 proteins. The most common therapeutic approaches include inhibition of S100 protein expression using microRNA-, small interfering RNA- or short hairpin RNA-based knockdown of S100 proteins using neutralizing antibodies or using specific small-molecule inhibitors. On the other side the role of CD4+ T cells (Th 17 cells) as a part of adaptive immunity, seems to be critical in the development of the skin lesions. Whether S100A7 or Th 17 cells are related to the severity of psoriasis is unclear. Immunohistology provides invaluable tools for better understanding psoriasis's pathogenetic mechanism and understanding the molecular processes involved in the pathogenesis of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* the study will include patients with psoriasis

Exclusion Criteria:

1. pregnancy
2. lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
immunohistochemical skin expression of S100A7 (psoriasin) | 1 year
  measuring the percentage area of S100A7 (psoriasin) positive cells in skin by immunohistochemistry
immunohistochemical skin expression of CD4 T cells | 1 year
  measuring number of CD4 T positive cells in skin by immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Iskandar IYK, Parisi R, Griffiths CEM, Ashcroft DM; Global Psoriasis Atlas. Systematic review examining changes over time and variation in the incidence and prevalence of psoriasis by age and gender. Br J Dermatol. 2021 Feb;184(2):243-258. doi: 10.1111/bjd.19169. Epub 2020 Jun 21. PMID 32358790
- [Background] Lowes MA, Suarez-Farinas M, Krueger JG. Immunology of psoriasis. Annu Rev Immunol. 2014;32:227-55. doi: 10.1146/annurev-immunol-032713-120225. PMID 24655295
- [Background] Yadav K, Singh D, Singh MR. Protein biomarker for psoriasis: A systematic review on their role in the pathomechanism, diagnosis, potential targets and treatment of psoriasis. Int J Biol Macromol. 2018 Oct 15;118(Pt B):1796-1810. doi: 10.1016/j.ijbiomac.2018.07.021. Epub 2018 Jul 11. PMID 30017989
- [Background] Michalek IM, Loring B, John SM. A systematic review of worldwide epidemiology of psoriasis. J Eur Acad Dermatol Venereol. 2017 Feb;31(2):205-212. doi: 10.1111/jdv.13854. Epub 2016 Aug 30. PMID 27573025